CLINICAL TRIAL: NCT07326579
Title: Effects of a Sleep Education Program Conducted by Occupational Health Nurse on the Health Status of Healthcare Workers Working 12-hour Alternating Day-night Shifts: a Multicentre Randomised Controlled Trial
Brief Title: Effects of a Sleep Education Program on the Health Status of Healthcare Workers Working 12-hour Alternating Day-night Shifts
Acronym: SLEEPMORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25PH236; 2025-A02584-45 (Other: N°ID RCB)
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers (HV)
Keywords: Sleep educational program; Alternating 12-hour; day and night shift

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep educational (Experimental): Personalized educational program
  Interventions: Behavioral: Sleep educational
- Control (No Intervention): Standard workplace medicine advice

INTERVENTIONS:
Behavioral: Sleep educational — Participants will undergo :
  * standardized monitoring initially (M0), then at 6 months (M6) and 12 months (M12)
  * a personalized educational program, including an initial consultation with a sleep doctor and a nurse, followed by monthly follow-ups with an occupational health nurse.
  Arms: Sleep educational

SUMMARY:
In a context of seeking a better balance between personal and professional life and labor shortages, the use of 12-hour alternating day-night shifts has become more common in work organizations, particularly in healthcare facilities. This work pattern combines exposure to alternating day and night shifts with long working hours, raising questions about its effects on health, particularly sleep quality and cardiovascular risk. Staff working alternating day/night or night shifts are at risk of cardiovascular disease, particularly in connection with sleep deprivation and the adoption of individual behaviors that increase the risk (smoking, poor diet, alcohol consumption, smoking and low physical activity). However sleep education is not integrated in a personalized way into the prevention advice provided by occupational health services.

Therefore, this study aims to investigate the effects of a 6-month sleep education program conducted by occupational health nursing staff, on the sleep duration of healthcare workers newly exposed to alternating 12-hour day and night shifts.

ELIGIBILITY:
Inclusion Criteria:

* Being a paramedical caregiverr (nurse or care assistant)
* Working 12-hour shifts (day/night)
* Working at least 80% of a full-time equivalent post
* Staff employed at a hospital listed among the investigating centers
* Being affiliated or entitled under a social security scheme
* Having received informed information about the study and have co- signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

* Nursing staff and nursing assistants who have been exposed for more than six months to alternating 12-hour shifts or atypical working hours (two eight-hour shifts, three eight-hour shifts or night shifts) during their professional career
* Nursing staff and nursing assistants with a history of mental illness or who are taking medication that affects alertness (psychotropic drugs)
* Pregnant or breastfeeding women
* Nursing staff or nursing assistants with sleep apnea syndrome, central hypersomnolence disorders, severe parasomnias, severe untreated restless legs syndrome
* Individuals with children under the age of 1 in the household
* Trans meridian travel (>2 time zones) during the month prior to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Effect of a 6-month sleep education program | 6 months
  Evaluate the effect of a 6-month sleep education program conducted by occupational health nursing staff on the sleep duration of nursing assistants newly exposed to alternating 12-hour day and night shifts.Absolute difference in average sleep duration (in minutes) measured over 14 days from an actigraph worn at the wrist, between Baseline (M0) and at 6 months (M6).

SECONDARY OUTCOMES:
Assess the impact of the sleep education program on sleep quality | 6 months
  The Pittsburgh Sleep Quality Index (PSQI) comprises 24 items, with scores ranging from 0 to 21, where a score > 5 indicates poor sleep quality)
Assess the impact of the sleep education program on participant state of health | 6 months
  Measure of cardiac frequency
Assess the impact of the sleep education program on quality of life | 6 months
  The Short Form 36 (SF-36) will be used to assess quality of life. This 36-item questionnaire includes 8 sub-scores ranging from 0 (minimum quality of life) to 100 (maximum well-being).
Assess the impact of the sleep education program on accidentology | 6 months
  Number of commuting accidents, workplace accidents, road accidents, near misses related to drowsiness

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Chu Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided